CLINICAL TRIAL: NCT00038870
Title: Therapy of Relapsed AML With Chemotherapy and Dendritic Cell Activated Lymphocytes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Immunex Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-075
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia
Keywords: AML; CML; Dendritic Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dendritic Cell Activated Lymphocytes (Experimental)
  Interventions: Biological: Dendritic Cell Activated Lymphocyte

INTERVENTIONS:
Biological: Dendritic Cell Activated Lymphocyte
  Other Names: autologous leukemia derived dendritic cell activated lymphocytes; DC/AL

SUMMARY:
1. Determine the feasibility of generation of autologous Acute Myelogenous Leukemia (AML) or Chronic Myelogenous Leukemia in myeloid blast crisis (CML/BC) derived dendritic cell activated lymphocytes (DC/AL) in poor prognosis patients.
2. Determine the toxicity of autologous leukemia derived dendritic cell activated lymphocytes (DC/AL) in patients with AML or CML/BC.
3. Quantitate circulating immune effector cells in patients after infusion of DC/AL.
4. Record the efficacy of AML or CML/BC derived dendritic cells and activated lymphocytes in promoting and sustaining remission in patients with AML or CML/BC.

DETAILED DESCRIPTION:
Most patients relapsing with AML either fail to achieve second remission or have only brief remissions. Patients more than 60 years of age or having histories of antecedent hematological disorders, prior chemotherapy, or poor risk cytogenetics have generally only short remissions and as a group have two year survivals of less than 10%. Equally patients with myeloid blast crisis of CML often fail to achieve remission or have responses of only brief duration. Laboratory studies have shown that AML leukemic blasts may be induced in culture to differentiate into dendritic cells which in turn may be used activate autologous lymphocytes to acquire leukemia specific cytotoxicity. This trial will assess the feasibility of generation of dendritic cell activated lymphocytes, and toxicity and efficacy of these activated cells given after reinduction chemotherapy. Before this study begins some toxicity information will have been generated in a trial of similar cells given to CML patients.

ELIGIBILITY:
Inclusion:

* AML patients either after first relapse or at diagnosis a) with high-risk cytogenetics such as -7, -5, +8, chromosome 9 or 11 abnormality, or b) WBC > 50,000, or c) age > 60 years*.
* AML patients are eligible for cell collection if they have > 1000 circulating blasts/mm at diagnosis.
* CML patients in myeloid blast crisis with > 1000 circulating blasts/mm.
* Creatinine <2, Bilirubin <3.
* Age >18.

Exclusion:

* Factors which would prevent the patient from receiving or cooperating with the full course of therapy or understanding the informed consent procedure.
* Concurrent or expected need for therapy with corticosteroids.
* Positive antibody to human immunodeficiency virus I.
* Acute promyelocytic Leukemia (FAB-M3).
* History of overt cardiac failure, systemic autoimmune disease or expected need for steroid therapy.

  * Patients >60 will be eligible for study but if found to have good prognosis cytogenetics (inversion (16) or t(8;21)) will subsequently be withdrawn from study and treated off protocol without infusion of autologous leukemia derived cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-01-31 (Actual); Primary Completion 2003-01-14 (Actual); Study Completion 2003-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Champlin, MD,BS, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org